CLINICAL TRIAL: NCT01975467
Title: CLAVICLE FRACTURE OUTCOMES: 1-3 YEAR FOLLOW UP OF DISPLACED MIDSHAFT FRACTURES TREATED WITH INTRAMEDULARY NAIL vs. NONOPERATIVE TREATMENT
Brief Title: Post Treatment Comparison Intramedullary Nail vs. Nonoperative Treatment
Status: Terminated | Type: Observational
Why Stopped: Low Enrollment
Sponsor: Sonoma Orthopedic Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRx-001
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Fracture of Clavicle
Keywords: midshaft clavicle fracture; intramedullary nail; sling
MeSH Terms: interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group - Nonoperative: Subjects that were treated with a sling for their displaced midshaft clavicle fracture.
- Test Group - Intramedullary Nail: Subjects that were treated with an intramedullary nail for their displaced midshaft clavicle fracture.
  Interventions: Device: CRx

INTERVENTIONS:
Device: CRx — The CRx is used to treat mid-shaft, with or without comminution clavicle fractures.
  Other Names: Intramedullary Nail
  Groups: Test Group - Intramedullary Nail

SUMMARY:
The objective of this post-market clinical study is to compare one to three year post treatment results, range of motion, strength, patient related functional outcomes and patient satisfaction, of internal fixation using the Sonoma Orthopedic Products CRx™ as compared to nonoperative management (e.g. sling) of similar displaced midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* A displaced transverse or oblique midshaft clavicle fracture with or without comminution
* Must be 12 ± 2 months to 36 ± 2 months post-treatment
* Must have received nonoperative treatment or operative treatment with a CRx™ device, no other devices, for their clavicle fracture
* Male or female at least 18 years of age
* Able to understand the requirements of the study, provide a written informed consent and comply with the study protocol
* Ability to understand and provide written authorization for use and disclosure of personal health information

Exclusion Criteria:

* Open, or segmental clavicle fracture
* Any clavicle or upper extremity fracture previous, concurrent, or subsequent to the study fracture
* Removal of the CRx™ device within 8 weeks of the study visit
* History of alcoholism
* Currently on chemotherapy or radiation therapy
* Habitual use of narcotic pain medications prior to injury or after injury for reasons other than clavicle pain
* Currently on worker's compensation
* History of a metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis
* Rheumatoid arthritis or other inflammatory arthropathies.
* History of chronic pain issues for reasons other than clavicle pain or psychiatric disorder that precludes reliable follow-up.
* Women that are pregnant or think that they might be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is open to anyone over the age of 18 that meet the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John LeBlanc, DO, Principal Investigator — North Coast Orthopaedics and Sports Medicine; Carl Basamania, MD, Principal Investigator — Madison Center/Polyclinic
Locations (2):
- United States (2):
  - North Coast Orthopaedics and Sports Medicine, Arcata, California
  - Madison Center/Polyclinic, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group - Nonoperative | Test Group - Intramedullary Nail
Started | 0 (Study terminated before enrollment) | 0 (Study terminated before enrollment)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group - Nonoperative | Test Group - Intramedullary Nail | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Gender
  Female |  |  | 0
  Male |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: DASH Score
Description: Subjects that are one to three years post-treatment will undergo an evaluation of fracture outcome utilizing the DASH instrument for function.
Time Frame: One time point
Population: Terminated due to low enrollment
Arm/Group | Control Group - Nonoperative | Test Group - Intramedullary Nail
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Range of Motion and Strength
Description: The ASES instrument will be used to assess range of motion and strength.
Time Frame: One time point
Arm/Group | Control Group - Nonoperative | Test Group - Intramedullary Nail
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group - Nonoperative | Test Group - Intramedullary Nail
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No